CLINICAL TRIAL: NCT06404853
Title: Multicenter Open-label Noncomparative Study to Evaluate the Effect and Safety of the Dietary Supplement Mannite in Pediatric Patients With Chronic Functional Constipation
Brief Title: Effect and Safety of the Dietary Supplement Mannite in Pediatric Patients With Chronic Functional Constipation
Acronym: MANNAPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: Iuppa Industriale S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASO.Ped.20.07
Record Dates: First submitted 2024-02-29; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Constipation - Functional
Keywords: constipation
MeSH Terms: conditions — Constipation | interventions — (1-6)-alpha-glucomannan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplement dietary manna (Other): Administration of supplement dietary manna
  Interventions: Dietary Supplement: Manna

INTERVENTIONS:
Dietary Supplement: Manna — Administration is by the oral route according to weight at a dosage of 1 g/kg/day, dissolved in a glass of water, up to a maximum of 30 g. Administration should be repeated every 24 h for 8 weeks, accompanied by plenty of hydration.
  In case an effective dosage is achieved (evacuation within 72 h) it will be maintained until the end of the study. If evacuation has not occurred after 72 h, evacuative enema and increased dosage to 1.5 g/kg/day will be indicated. If further evacuative enema is needed, product administration will be discontinued and classical polyethylene glycol therapy will be started as per guidelines.

SUMMARY:
Functional constipation is a widely prevalent pediatric issue, with a prevalence in some studies as high as 32.2%.

Treatment consists of a combination of behavioral and pharmacological interventions (mainly, administration of polyethylene glycol laxatives or the use of enemas).

Glucomannan (GNN) is a polysaccharide of 1,4-D-glucose and D-mannose found in the soluble fiber of some plants. While studies available in the literature to date agree that mannite is a dietary supplement with safe use, the usefulness of this compound remains controversial.

DETAILED DESCRIPTION:
Functional constipation is a widely prevalent pediatric issue, with a prevalence in some studies as high as 32.2%. Characterized by annoying and embarrassing symptoms such as reduced number of evacuations, increased stool consistency, fecal incontinence, and abdominal pain functional constipation has a negative impact on the quality of life of affected children and their families. It is a frequent reason for referral to the general pediatrician and pediatric gastroenterologist and significantly impacts health care spending The guidelines publicized by the European Society for Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) and the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN) on functional constipation in children provide the most up-to-date evidence-based recommendations for the evaluation, treatment and follow-up of children with this condition. Key indications include a diagnosis based on history and physical examination and a definition of functional constipation based on the criteria of Rome.

Treatment consists of a combination of behavioral and pharmacological interventions (mainly, administration of polyethylene glycol laxatives or the use of enemas).

Glucomannan (GNN) is a polysaccharide of 1,4-D-glucose and D-mannose found in the soluble fiber of some plants. While studies available in the literature to date agree that mannite is a dietary supplement with safe use, the usefulness of this compound remains controversial.

The study aims to evaluate the effect of Mannite supplement (composed of 90% Mannite from Fructose and 10% Manna from Ash) as a unique therapy in the treatment of functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of functional constipation defined according to Rome IV criteria.
* Age between 6 months and 16 years.
* Informed consent signed by parent/legal guardian

Exclusion Criteria:

* Presence of organic causes of bowel disorders (Hirschsprung's disease, spinal abnormalities or anorectal pathology; history of gastro-intestinal surgery), celiac disease
* Mental retardation
* Irritable bowel syndrome
* Taking medications that affect gastro-intestinal motility in the previous 4 weeks
* Clinical suggestive of metabolic disease (e.g., hypothyroidism)
* Known hypersensitivity to manna, mannitol, or other ingredient in the dietary supplement mannite

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Outcome of therapeutic effect | At 8 weeks
  The therapeutic outcome assessment of the mannitol-based dietary supplement in the treatment of pediatric constipation will be evaluated through the following endpoint:
  · Spontaneous bowel movements more than twice per week.
Outcome of therapeutic effect | At 8 weeks
  The therapeutic outcome assessment of the mannitol-based dietary supplement in the treatment of pediatric constipation will be evaluated through the following endpoint:
  · Absence of soiling episodes.
Outcome of therapeutic effect | At 8 weeks
  The therapeutic outcome assessment of the mannitol-based dietary supplement in the treatment of pediatric constipation will be evaluated through the following endpoint:
  · Number of painful evacuations or evacuations with hard stools per week.
Outcome of therapeutic effect | At 8 weeks
  The therapeutic outcome assessment of the mannitol-based dietary supplement in the treatment of pediatric constipation will be evaluated through the following endpoint:
  · Number of episodes of abdominal pain per week.
Outcome of therapeutic effect | At 8 weeks
  The therapeutic outcome assessment of the mannitol-based dietary supplement in the treatment of pediatric constipation will be evaluated through the following endpoint:
  · Need for evacuative enema treatment due to lack of evacuation for three consecutive days.
Outcome of therapeutic effect | At 8 weeks
  The therapeutic outcome assessment of the mannitol-based dietary supplement in the treatment of pediatric constipation will be evaluated through the following endpoint:
  · Number of flatulence episodes within a week.

SECONDARY OUTCOMES:
Outcome of safety | At 8 weeks
  The safety outcome assessment of the mannitol-based dietary supplement in the treatment of pediatric constipation will be evaluated through the following endpoints:
  * Absence of gastrointestinal-related adverse events during the study period.
  * Other adverse events (mild or severe) reported by parents during the study period, including pain, infections, or any other events related to the intervention
Questionnaire Pediatric Quality of Life Inventory Gastrointestinal Symptoms Module | Every week for 8 weeks
  The questionnaire PedsQL Gastrointestinal Symptoms Module has a scale that typically ranges from 0 to 100: higher scores indicate a better outcome, representing fewer symptoms and higher health-related quality of life.
Number of Bowel Movements | Daily for 8 weeks
  Number of bowel movements, recorded daily
Stool Consistency | Daily for 8 weeks
  Daily dairy of stool consistency, assessed using the Bristol Stool Scale, which categorizes stool types from 1 "very costipated" to 7 "Inflammation and Diarrhea".
Involuntary Fecal Loss | Daily for 8 weeks
  Daily dairy of involuntary fecal loss with Yes/No indicator.
Additional Symptoms | Daily for 8 weeks
  Daily dairy of additional symptoms such as bloating (sensation of a swollen belly), abdominal pain, discomfort (general abdominal disturbance), and straining during defecation

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Felici, Principal Investigator — Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo
Locations (1):
- SC Pediatria, Alessandria, Piedmont, Italy